CLINICAL TRIAL: NCT00336921
Title: A Double-blind, Randomized,Placebo Controlled Study of Alfuzosin 10mg od in the Return to Successful Voiding in Patients With a First Episode of Acute Urinary Retention Due to Benign Prostatic Hyperplasia
Brief Title: Alfuzosin for Treating Acute Urinary Retention
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Sanofi (Industry)
Responsible Party: Medical Affairs Study Director, sanofi-aventis
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: L_9645
Record Dates: First submitted 2006-06-14; First posted 2006-06-15 (Estimated); Last update posted 2009-09-15 (Estimated); Status verified 2009-09

CONDITIONS: Acute Urinary Retention
MeSH Terms: interventions — alfuzosin

ARMS (2):
- 1 (Active Comparator): Alfuzosin 10mg
  Interventions: Drug: Alfuzosin
- 2 (Placebo Comparator): Placebo
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Alfuzosin — Once daily
  Arms: 1
Drug: Placebo — Once daily
  Arms: 2

SUMMARY:
The primary objective of the study is to assess the efficacy of alfuzosin 10mg daily in the return to successful voiding after removal of the catheter following a first episode of acute urinary retention (AUR) in patients suffering from benign prostatic hyperplasia (BPH).

ELIGIBILITY:
Inclusion Criteria:

* First episode of painful AUR related to BPH requiring catheterization
* Residual volume between 500ml and 1500ml obtained at the time of catheterization and during the first one hour after catheterization

Exclusion Criteria:

* Participated in another investigational study within 3 months before recruitment
* Suspect bladder neuro-dysfunction unrelated to etiology;
* Single Bladder neck disease;
* Acute/chronic prostatitis;
* Diagnosed prostate carcinoma;
* Suspected prostate carcinoma diagnosed by ultrasound wave;
* Surgical history of prostate and urethra;
* Diagnosed/suspected abnormality in urethra structure;
* Bladder stone;
* Blood urine retention caused by any reason;
* Residual volume less than 500 ml
* Residual volume more than 1500 ml
* AUR not due to BPH
* Parkinson's disease
* Insulin dependent diabetes
* Known/suspected multiple sclerosis;
* Stroke/MI within 6 months prior to enrolment;
* AST, ALT and Creatinine > 1.5x upper limit; neutrophil < 3,000/mm³; platelet < 100,000/mm³;
* Unstable/severe heart failure;
* History of postural hypertension/hypotension;
* Known hypersensitivity to α-receptor blocker;
* Suspected/diagnosed expansible nerval disease;
* Treatment with sympathomimetic agent within 1 week prior to enrolment, except OTC drug for cold intermittently;
* Treatment with α1-receptor blocker within 1 month prior to enrolment;
* Treatment with tricyclic antidepressants, anticholinergic agents, sympathomimetic agent (other than the above reason), first generation antihistaminic, except the treatment with stable β sympathomimetic agent/ anticholinergic agents lasting more than 1 week for Asthma and COPD (Chronic Obstructive Pulmonary Disease);
* Treatment with Disopyramide

The above information is not intended to contain all considerations relevant to a patient's potential participation in a clinical trial.

Ages: 50 Years to 80 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 156 (Actual)
Dates: Start 2006-02; Primary Completion 2007-04 (Actual)

PRIMARY OUTCOMES:
Percentage of patients with successful voiding after catheter removal | Day 3 and 4
Adverse events | From the beginning to the end of the study

CONTACTS AND LOCATIONS:
Overall Officials: Bruno Jolain, Study Director — Sanofi
Locations (1):
- Sanofi-aventis, Beijing, China